CLINICAL TRIAL: NCT02226731
Title: Assessment of the Efficacy of Early Intrauterine Tamponade With a Belfort-Dildy Balloon Obstetric Tamponade System in the Treatment of Immediate Postpartum Hemorrhage
Brief Title: Intrauterine Tamponade With a Belfort-Dildy Balloon in the Treatment of Immediate Postpartum Hemorrhage
Acronym: TUB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P130914
Record Dates: First submitted 2014-08-06; First posted 2014-08-27 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Immediate Postpartum Hemorrhage
Keywords: Immediate postpartum hemorrhage; Intrauterine balloon tamponade
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Belfort-Dildy balloon device (Experimental)
  Interventions: Device: Early Belfort-Dildy Balloon
- Late Belfort-Dildy balloon device (Other)
  Interventions: Device: Late Belfort-Dildy balloon

INTERVENTIONS:
Device: Early Belfort-Dildy Balloon — Intrauterine tamponade with the Belfort-Dildy balloon, performed in the 15 minutes after randomization at the same time as the second line uterotonic treatment.
  Arms: Early Belfort-Dildy balloon device
Device: Late Belfort-Dildy balloon — Intrauterine tamponade with the Belfort-Dildy balloon, performed if failure of second line uterotonic treatment, ie persisting bleeding 30 minutes after the beginning of this infusion.
  Arms: Late Belfort-Dildy balloon device

SUMMARY:
The purpose of this study is to evaluate the impact of early intrauterine tamponade with a Belfort-Dildy balloon catheter in immediate postpartum hemorrhage(IPPH) after vaginal delivery and refractory to first-line uterotonic treatment, ie performed at the same time as second line uterotonic treatment, as compared tolate intrauterine tamponade performed in case of failure of second line uterotonic treatment, on the final severity of PPH. ).

DETAILED DESCRIPTION:
Immediate postpartum hemorrhage (IPPH) is among the most frequent causes of pregnancy-related mortality in both the USA and in Europe. In France, IPPH remains the leading cause of maternal mortality, responsible for 18% of the maternal deaths and 90% of the deaths from IPPH are considered avoidable. The initial treatment of severe IPPH involves medical management, uterine massage, and uterotonic drugs such as oxytocin, ergometrine, and prostaglandins or their analogues; In France oxytocin is used as the first line uterotonic, and Sulprostone as the second line uterotonic. When these first-line medical treatments fail, invasive therapies, including uterine compression suture, pelvic vascular ligation, or arterial embolization can be used, individually or in combination. Hysterectomy is the ultimate measure to control a hemorrhage and save the mother's life. Nonetheless, the management of severe IPPH is less well standardized than its prevention, especially after the failure of uterotonic drugs, as demonstrated by the heterogeneity of practices between countries and even between hospitals in the same country. These invasive treatments require specific and expensive technical and human resources and have adverse effects. That is why, over the last years, intra-uterine tamponade with balloon has been increasingly used; indeed, it is a new minimally invasive method that can be used directly in the delivery room, at the initial stage of second-line treatments; it could accelerate the control of IPPH, limit recourse to these surgical or interventional radiology treatments, and reduce the quantity of blood products transfused. Intrauterine balloon tamponade thus appears to be a potentially additional effective strategy for obtaining hemostasis in the case of IPPH refractory to conventional uterotonic treatments. Despite the fact that the current literature assessing its efficacy is limited to case series and before-after observational studies, the available evidence suggests that it is associated with a drop in the need for invasive treatments. Based on this evidence, intra-uterine tamponade balloon has been included in guidelines for PPH treatment in many countries, including France, and it has widely spread in clinical practices. The clinical question that is now arising is its optimal timing in the management of PPH. It is currently classically performed after failure of second-line uterotonic treatment but it is possible that its earlier use, after failure of first-line uterotonic treatment, could further decrease the rate of severe PPH.

A randomized controlled trial is therefore necessary to determine the optimal timing of intrauterine balloon tamponade in the treatment of PPH. .

We propose a multicenter, randomized open treatment trial with two parallel arms. The trial will be conducted in 21 maternity units. Before inclusions begin, the medical staff will be trained in the use of the obstetric tamponade system to be used in the trial. For each woman with IPPH refractory to first line uterotonic, the eligibility criteria will be immediately verified, the woman informed and her written informed consent obtained if that is possible. If not, the woman can nonetheless be randomized and she will be secondarily informed and her consent requested. The randomization list will be centralized and generated by a computer program under the supervision of the Paris Centre Clinical Research Unit. Allocation to a study arm will be performed on a secure Internet platform (CleanWeb) always accessible (24/7) in each delivery room. The clinician including the patient will know her allocation immediately.

The management of randomized women will depend on the arm to which they are allocated:

* In the Experimental arm : the intravenous second line uterotonic Sulprostone infusion will be immediately combined with an intrauterine tamponade with the Belfort-Dildy balloon. Balloon insertion and inflation will follow a standardized protocol. Its intrauterine position will be verified by abdominal ultrasound. If the bleeding persists from the cervix or the balloon catheter drainage port 30 minutes after the beginning of the Sulprostone infusion, the tamponade will be considered a failure and an invasive emergency procedure by interventional radiology or surgery will be arranged and performed immediately after the removal of the balloon in the operating room.
* In the Control arm, women will only receive the Sulprostone infusion first. If bleeding persists 30 minutes after the beginning of this infusion, an intrauterine tamponade with the Belfort-Dildy balloon will be performed. Balloon insertion and inflation will be performed following the standardized protocol. If the bleeding persists from the cervix or the balloon catheter drainage port 15 to 30 minutes after the introduction of the balloon, the tamponade will be considered a failure and an invasive emergency procedure by interventional radiology or surgery will be arranged and performed immediately after the removal of the balloon in the operating room.

In both arms, all patients will have an indwelling urinary catheter and will receive antibiotic prophylaxis (amoxicillin-clavulanic acid and gentamicin) beginning with the Sulprostone infusion and continuing for 48 hours. The other components of IPPH management (fluid resuscitation, transfusion, resuscitation) will comply with national guidelines. If the bleeding stops, the patient will be transferred to a continuous care or post-interventional monitoring unit. Monitoring will be conducted by the investigator who included the patient. A venous blood sample will be collected on the 2nd day postpartum to measure hemoglobin and hematocrit values. The data will be entered as they are collected throughout the trial with Cleanweb software.

The duration of the participation of each patient included in the trial will be from inclusion through postpartum visit, or a maximum of approximately 8 weeks after the delivery. The maximum duration of study treatment will be 24 hours for each patient included in the protocol.

The total duration of the trial will be 36 months including 24 months of patient inclusion: the first 4 months, before the beginning of the inclusion period will be devoted to training staff in the use of the balloon tamponade system and in compliance with the trial protocol and the 8 months following the end of the inclusion period will be used to finalize the data collection, clean the database and analyze it.

ELIGIBILITY:
Inclusion Criteria:

The trial will include women:

* aged 18 years or older,
* who have just had a vaginal delivery
* between 35 and 42 weeks of gestation
* with a PPH persisting 15 minutes after the injection of 5 UI or 10 IU of oxytocin by slow IV and uterine massage,
* and who provided informed written consent. If her condition does not allow her consent to be obtained immediately in ethically acceptable conditions, it may be obtained from her healthcare agent, or if there is none, from a family member, if present. In case where neither a healthcare agent nor a family member is present on the day of inclusion, the patient can nonetheless be included. She will be informed secondarily, and her consent will be requested for the potential continuation of the research and use of her data
* Patient beneficiary or affiliated to a health insurance

Exclusion Criteria:

The trial will not include women:

* who have just had a cesarean delivery
* with a contraindication to Sulprostone
* with clinical chorioamnionitis or an in utero fetal death
* or a medically-indicated termination of pregnancy
* with PPH secondary to cervicovaginal lacerations without any uterine hemorrhage, uterine rupture, or placenta accreta
* with arterial bleeding requiring embolization
* with a purulent infection of the cervix, vagina or uterus
* with symptoms indicating a hysterectomy
* with cervical cancer
* with a uterine malformation
* or who refuses to sign the informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Proportion of women who received at least 3 RBC units for the treatment of PPH and /or who had a calculated peripartum blood loss > 1000 ml. | 1 day
  With Calculated peripartum blood loss= estimated blood volume × ((prepartum Ht - Day 2postpartum Ht)/prepartum Ht ) and Estimated blood volume (ml) = booking weight (kg) × 85)

SECONDARY OUTCOMES:
Other markers of severe hemorrhage | 1 day
  Incidence of each component of the primary outcome
Other markers of severe hemorrhage | 24 hours
  Proportion of women with a total blood loss in the first 24 hours postpartum ≥ 1500 mL (estimated or measured).
Other markers of severe hemorrhage | 8 days
  Proportion of women receiving a postpartum RBC transfusion
Other markers of severe hemorrhage | 8 days
  Mean number of units of packed red blood cells transfused in postpartum
Other markers of severe hemorrhage | 8 days
  Proportion of women receiving at least 4 units of packed red blood cells.
Other markers of severe hemorrhage | 2 days
  Proportion of women with a difference ≥ 4 g/dL between the hemoglobin value before and on the 2nd day after delivery in the absence of a transfusion of packed red blood cells.
Other markers of severe hemorrhage | 2 days
  Mean difference between the hemoglobin values before delivery and on the 2nd day postpartum in the absence of a transfusion of packed red blood cells.
Other markers of severe hemorrhage | 2 days
  Mean difference between the hematocrit values before delivery and on the 2nd day postpartum in the absence of a transfusion of packed red blood cells
  .
Other markers of severe hemorrhage | 2 days
  Total calculated peripartum blood loss
  .
Other markers of severe hemorrhage | 2 days
  Proportion of women with a total calculated peripartum blood loss ≥ 1500 mL
  .
Other markers of severe hemorrhage | 2 days
  Proportion of women transferred to Intensive care unit
Other markers of severe hemorrhage | 1 day
  Proportion of women who had invasive second line therapy, any of the following : arterial embolization, pelvic arterial ligation, uterine compression suture, hysterectomy
other Genital tract infection | 8 days
  Assessed by :
  * Proportion of women with a temperature >38°5C during postpartum hospitalization
other Genital tract infection | 8 days
  Assessed by :
  * Proportion of women with endometritis during postpartum hospitalization.
other Genital tract infection | 6 weeks
  Assessed by :
  • Proportion of women who had endometritis at the 6 weeks postpartum visit.
Other markers of severe hemorrhage | 24 hours
  Proportion of women with a total blood loss in the first 24 hours postpartum ≥ 2000 mL (estimated or measured)
Other markers of severe hemorrhage | 2 days
  Proportion of women with a total calculated peripartum blood loss ≥ 2000 mL

CONTACTS AND LOCATIONS:
Overall Officials: Patrick ROZENBERG, MD, Principal Investigator — Department of Obstetrics, Poissy-Saint Germain Hospital Center; Catherine DENEUX - THARAUX, MD, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- CHI de Poissy Saint Germain en Laye, Poissy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rozenberg P, Sentilhes L, Goffinet F, Vayssiere C, Senat MV, Haddad B, Morel O, Garabedian C, Vivanti A, Perrotin F, Kayem G, Azria E, Raynal P, Verspyck E, Sananes N, Gallot D, Bretelle F, Seco A, Winer N, Deneux-Tharaux C; Groupe de Recherche en Obstetrique et Gynecologie. Efficacy of early intrauterine balloon tamponade for immediate postpartum hemorrhage after vaginal delivery: a randomized clinical trial. Am J Obstet Gynecol. 2023 Nov;229(5):542.e1-542.e14. doi: 10.1016/j.ajog.2023.05.014. Epub 2023 May 18. PMID 37209893
- [Background] Laas E, Bui C, Popowski T, Mbaku OM, Rozenberg P. Trends in the rate of invasive procedures after the addition of the intrauterine tamponade test to a protocol for management of severe postpartum hemorrhage. Am J Obstet Gynecol. 2012 Oct;207(4):281.e1-7. doi: 10.1016/j.ajog.2012.08.028. Epub 2012 Aug 17. PMID 23021688
- [Background] Georgiou C. Balloon tamponade in the management of postpartum haemorrhage: a review. BJOG. 2009 May;116(6):748-57. doi: 10.1111/j.1471-0528.2009.02113.x. PMID 19432563
- [Background] Tindell K, Garfinkel R, Abu-Haydar E, Ahn R, Burke TF, Conn K, Eckardt M. Uterine balloon tamponade for the treatment of postpartum haemorrhage in resource-poor settings: a systematic review. BJOG. 2013 Jan;120(1):5-14. doi: 10.1111/j.1471-0528.2012.03454.x. Epub 2012 Aug 13. PMID 22882240
- [Background] Revert M, Cottenet J, Raynal P, Cibot E, Quantin C, Rozenberg P. Intrauterine balloon tamponade for management of severe postpartum haemorrhage in a perinatal network: a prospective cohort study. BJOG. 2017 Jul;124(8):1255-1262. doi: 10.1111/1471-0528.14382. Epub 2016 Oct 25. PMID 27781401
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374